CLINICAL TRIAL: NCT04707105
Title: A Prospective Observational Cohort Study in Chinese Patients With Primary Intracerebral Hemorrhage
Brief Title: Prospective Cohort Study of Intracerebral Hemorrhage
Acronym: POSTER
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2018001098
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: primary intracerebral hemorrhage; hypertension; perihematomal edema; secondary brain injury; remote diffusion-weighted imaging lesions (R-DWILs); immune response; multimodel image; cohort; MRI
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Second Affiliated Hospital, School of Medicine, Zhejiang University: a prospective cohort of patients of primary intracerebral hemorrhage in Second Affiliated Hospital, School of Medicine, Zhejiang University
- Second People's Hospital of Hangzhou City, Zhejiang Province: a prospective cohort of patients of primary intracerebral hemorrhage in Second People's Hospital of Hangzhou City, Zhejiang Province
- 4th Affiliated Hospital, School of Medicine at Zhejiang University: a prospective cohort of patients of primary intracerebral hemorrhage in 4th Affiliated Hospital, School of Medicine at Zhejiang University

SUMMARY:
The investigators design a prospective, observational cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective ,treatments and prognosis of Chinese hospitalised adult patients with intracerebral hemorrhage.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) remains a devastating disease with high mortality, yet few therapeutic managements have been proved effective. Large quantities of work needs to be done to fully delineate the prevalence and prognosis of ICH. Hence, the investigators design a prospective, observational cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective, treatments and prognosis of Chinese hospitalised adult patients with ICH.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients over 18 years old of primary intracerebral hemorrhage.

Exclusion Criteria:

1. patients of secondary intracerebral hemorrhage，such as hemorrhagic transformation of ischemic stroke, aneurysmal, cavernomas, arterio- venous malformations, central venous thrombosis, trauma-related, or tumor.
2. isolated intraventricular hemorrhage or subarachnoid hemorrhage pregnant patients；
3. surgical evacuation of hematoma；
4. unavailability to get complete blood cell samples and presenting contraindications or refusal to MRI
5. patients cannot be followed up for any reasons.
6. patients death in 24 hours
7. pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 856 hospitalized patients over 18 years old with primary intrcerebral hemorrhage will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 856 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with a 3-month modified Rankin Scale (mRS) score≤ 3 | 2-3years
  mRS 0-6, higher indicate worse outcome

SECONDARY OUTCOMES:
Absolute peripheral hematoma edema(PHE) growth | 2-3years
  absolute peripheral hematoma edema growth in CT/MRI measured by picture archiving and communication systems(PACS) system
Relative peripheral hematoma edema(rPHE) | 2-3years
  rPHE：absolute PHE divided by hematoma volume in CT/MRI
National institute of health stroke scale（NIHSS score） | 2-3years
  NIHSS 0-42, higher indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, MD,PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided